CLINICAL TRIAL: NCT02691234
Title: Safety and Efficacy of Low Intensity Shockwave Therapy in Treating Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0592-HMO-CTIL
Record Dates: First submitted 2016-01-31; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Extracorporeal Shockwave Therapy; Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extracorporeal Shockwave Therapy and debridement (Experimental): The treatment will be performed as an outpatient care procedure with no anesthesia. Patients will undergo wound debridement and cleansing before each treatment. The transducer device will be positioned against the lesion area and shockwaves will be delivered at a gradually increasing energy, with a maximum energy level of 0.09mJ/mm2
  Interventions: Device: Extracorporeal Shockwave Therapy and debridement; Other: debridement and cleaning
- debridement and cleansing. (Active Comparator): The standard treatment to the control group and the treatment group will be performed as an outpatient care procedure with no anesthesia. Patients will undergo wound debridement and cleansing. The physician will treat the patient in regard to his medical state: antibiotic medication if needed, dressing and off loading with Orthotic devices
  Interventions: Other: debridement and cleaning

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy and debridement
  Arms: Extracorporeal Shockwave Therapy and debridement
Other: debridement and cleaning

SUMMARY:
Low intensity shockwaves for treating diabetic foot ulcers (DFUs) have been in evaluation for the past 5 years. Many researchers showed the effectiveness of Low intensity shockwaves of in accelerating the healing rate of non-ischemic chronic DFUs. Wang et al. showed, the use of Low intensity shockwaves on DFUs, significantly improved topical blood flow perfusion rate, increased cell proliferation and cell activity and decreased cell apoptosis.

The present study deals with the effect of low intensity shockwaves on DFUs. Shockwave treatment will be done together with the standard conventional treatment for DFUs, compared to a control group who will receive the same conventional standard of care.

ELIGIBILITY:
* Inclusion Criteria:

  1. Chronic non-healing diabetic foot ulcers for more than 2 months.
  2. Age 18-80 years
  3. Ankle Brachial Index (ABI) ≥0.6
  4. Diabetic Foot Ulcer with the long diameter of ≤7cm and a short diameter of ≥1cm
  5. The target ulcer is up to Wagner's grade 3
  6. Albumin level ≥25g/L
  7. Hemoglobin level ≥90g/L
  8. Estimated Glomerular Filtration Rate (eGFR) ≥30ml/min/1.73m2
  9. The patient agrees to comply with study protocol requirements, including the shockwave procedure, self-care of the ulcer (dressings, orthotics etc.) and all follow-up visit requirements
* Exclusion Criteria:

  1. Pregnancy or lactation
  2. ABI <0.6
  3. The long diameter of the target ulcer is >7cm and the short diameter is <1cm
  4. The target ulcer is of Wagner's grade 4 or above
  5. Severe Hypoalbuminemia <25g/L
  6. Severe anemia, Hemoglobin level <90g/L
  7. eGFR <30ml/min/1.73m2
  8. Patients suffering from acute Charcot foot
  9. Severe edema of the treated limb
  10. Patient with present malignancy or past malignancy in the treated area
  11. Systemic chemotherapy/ radiation treatment within the last 6 months
  12. Deep vein thrombosis within the last 6 months
  13. Any other experimental treatment or participation in other studies

      -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
To assess initial closure rate of the wound 4 weeks after the last treatment session, as compared to the control group receiving conventional standard of care. | four weeks

IPD SHARING:
Plan to Share IPD: No